CLINICAL TRIAL: NCT05269342
Title: Nurse-led Exercise To Improve Shoulder Pain, Shoulder Disability, and Quality of Life in Postoperative Patients With Newly Diagnosed Head and Neck Cancer
Brief Title: Nurse-led Exercise Improves Shoulder Pain, Shoulder Disability, and Quality of Life in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YU LONG HONG (Other)
Responsible Party: Sponsor-Investigator, YU LONG HONG, Principal Investigator, Hualien Tzu Chi General Hospital
Organization: Hualien Tzu Chi General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HYL
Record Dates: First submitted 2022-02-18; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Cancer; Cancer of Head and Neck; Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the nurse-led counseling and after intervention exercise (Experimental): The NUCAI aims to help patients manage themselves physically and psychologically by giving support, education, and exercise tracking.
  The participants in the control group were care as usual.Intervention group were the nurse-led counseling and after intervention exercise (NUCAI), in patients with HNC.
  Interventions: Behavioral: nurse-led counseling and after intervention

INTERVENTIONS:
Behavioral: nurse-led counseling and after intervention — the nurse-led counseling and after intervention exercise (NUCAI), in patients with HNC

SUMMARY:
Background: This study aimed to the postoperative patients with newly diagnosed head and neck Cancer. The nurse-led counselling and after intervention improved shoulder pain, Shoulder Disability, and Quality of Life., before 2 weeks radical neck dissection and at postoperative 2, 4, 8, and 12 weeks.

Methods：Participants were identified for eligibility from the otorhinolaryngology outpatient department of a medical center in eastern Taiwan. The data of 40 patients were collected between Aug 1, 2017, and Jul 31, 2018. 40 participants were randomly assigned to an experimental (n = 20) and a control group (n = 20). The experimental group received the nurse counselling and after intervention exercise intervention , and the control group received usual care. Study tools used were the shoulder pain and disability indices, University of Washington Quality of Life Questionnaire.

DETAILED DESCRIPTION:
Head and neck cancer (HNCs) is malignancies . Globally, HNCs was the seventh most common cancer in 2018. In taiwan, have high incidences . Primary treatments for HNCs are surgery alone or in combination with radiation . The radical neck dissection and radiotherapy inevitably damage nerves and muscles, resulting in various complications such as shoulder pain and disability; the shoulder disability and chronic neck pain occur following radical neck dissection, these complications may considerably limit the individual's capacity to undertake various tasks, affecting daily physical activities. Immediate postoperative rehabilitation has been advocated to improve these complications in HNC participants . But rticipants often fail to achieve this thresh old, which emphasizes the need to change their inactive behaviour.

Nurses are involved in patient care and have the necessary skills and knowledge about the medical and practical aspects of head and neck cancer treatment . Nurses can provide information, support and coaching to HNC participants .Nurses are in a key position to deliver an intervention to improve QoL . The investigators designed a randomised controlled trial (RCT) to investigate the effectiveness of a comprehensive 12weeks nurse-led intervention, the nurse counselling and after intervention (NUCAI), in HNC participants follow exercise intervention

ELIGIBILITY:
Inclusion Criteria:

aged >20 years old newly diagnosed with HNC scheduled to receive surgery had no serious complications had no history of mental illness had no comorbidities had no sensory-cognitive problems could understand Chinese or Taiwanese

Exclusion criteria:

could not communicate or comprehend the questionnaires had a history of shoulder dysfunction before neck dissection had preexisting shoulder pain, dysfunction, or weakness had any disorders that could influence movement performance.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-09-09 (Actual)

PRIMARY OUTCOMES:
Demographic and Illness-related Information | 2 weeks preoperatively
  age, sex, educational level, and cancer stage

SECONDARY OUTCOMES:
shoulder pain and disability indices | 2 weeks preoperatively (baseline) and then 2, 4, 8, and 12 weeks postoperatively
  shoulder pain and disability

OTHER OUTCOMES:
the University of Washington Quality of Life Questionnaire (UW-QOL) | 2 weeks preoperatively (baseline) and then 2, 4, 8, and 12 weeks postoperatively
  Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Yu Long Hong, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No